CLINICAL TRIAL: NCT03251300
Title: Mirabegron for Female Patients With Overactive Bladder Syndrome: Comparison of Daytime and Nighttime Dosing
Brief Title: Mirabegron for Female OAB Patients: Comparison of Daytime and Nighttime Dosing
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 106001-F
Record Dates: First submitted 2017-08-10; First posted 2017-08-16 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Overactive Bladder Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): daytime dosing of mirabegron
  Interventions: Drug: daytime dosing of mirabegron
- group B (Active Comparator): nighttime dosing of mirabegron
  Interventions: Drug: nighttime dosing of mirabegron

INTERVENTIONS:
Drug: daytime dosing of mirabegron — All OAB female patients will receive daytime dosing (08:00 AM) of mirabegron
  Arms: group A
Drug: nighttime dosing of mirabegron — All OAB female patients will receive nighttime dosing (08:00 PM) of mirabegron
  Arms: group B

SUMMARY:
The aim of this study is to elucidate whether night-time dosing of mirebegron can improve nocturia, compared with daytime dosing of mirabegron.

DETAILED DESCRIPTION:
Background/Purpose: Women with overactive bladder syndrome (OAB) may have symptoms of nocturia, in addition to urgency and frequency. Women with nocturia are prone to suffer from a fall and fracture. Beta-3 agonist is an effective treatment for OAB. However, women with nocturia may need adjuvant desmopressin to improve nocturia. The aim of this study is to elucidate whether night-time dosing can improve nocturia, compared with daytime dosing.

Patients and Methods: The investigators will perform a prospective randomized controlled trial to recruit 90 female OAB patients at the outpatient clinic of Department of Obstetrics and Gynecology of Far Eastern Memorial Hospital. All OAB women will be treated by mirabegron. All enrolled OAB women will be allocated to two groups (group A and B). The women in group A will receive daytime dosing of mirabegron treatment; and the women in group B will receive nighttime dosing of mirabegron. All OAB female patients will be asked to complete Urgency Severity Scales, Overactive Bladder Symptoms Scores questionnaires, King's Health questionnaires, 3-day bladder diary before, 4 weeks' and after 12 weeks' mirabegron treatment. STATA software is used for statistical analyses.

Possible Results: The investigators can answer whether night-time dosing of mirabegron can improve nocturia, compared with daytime dosing.

ELIGIBILITY:
Inclusion Criteria:

* OAB symptoms for at least one month
* >20 years

Exclusion Criteria:

* Allergy to mirabegron, urinary tract infections, unstable hypertension

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Nocturia episodes | 12 weeks
  comparison of baseline and post-treatment nocturia episodes from bladder diary

SECONDARY OUTCOMES:
Severity of nocturia | 12 weeks
  comparison of baseline and post-treatment severity of nocturia from questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

REFERENCES:
- [Result] Tsai KH, Hsiao SM, Lin HH. Tolterodine treatment of women with overactive bladder syndrome: Comparison of night-time and daytime dosing for nocturia. J Obstet Gynaecol Res. 2017 Nov;43(11):1719-1725. doi: 10.1111/jog.13438. Epub 2017 Jul 16. PMID 28714288
- [Derived] Hsiao SM. Mirabegron nighttime versus daytime dosing for women with overactive bladder syndrome: a randomized controlled trial. Sci Rep. 2025 Aug 21;15(1):30687. doi: 10.1038/s41598-025-15780-5. PMID 40841399